CLINICAL TRIAL: NCT02518217
Title: ShapeUp Empower Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Rena R. Wing, Professor, Director of the Weight Control and Diabetes Research Center, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShapeUpEmpower2015
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Apps Only (Active Comparator)
  Interventions: Behavioral: Weight Loss Apps
- ShapeUp Empower (Experimental)
  Interventions: Behavioral: Weight Loss Apps; Behavioral: ShapeUp Empower
- ShapeUp Empower + Incentives (Experimental)
  Interventions: Behavioral: Weight Loss Apps; Behavioral: ShapeUp Empower; Behavioral: Financial Incentives for Engagement

INTERVENTIONS:
Behavioral: Weight Loss Apps — Provision of commercially available smartphone applications for healthy eating, physical activity, and weight loss.
Behavioral: ShapeUp Empower — Online intervention with training in behavioral strategies for healthy eating, physical activity, and weight loss. Includes periodic feedback on weight loss progress and engagement with the intervention platform.
  Arms: ShapeUp Empower; ShapeUp Empower + Incentives
Behavioral: Financial Incentives for Engagement — Financial incentives for completing tasks such as viewing instructional information and reporting self-monitored body weights via the study website.
  Arms: ShapeUp Empower + Incentives

SUMMARY:
This randomized controlled trial will evaluate patterns of use and health outcomes of the ShapeUp Empower online program with and without financial incentives for program engagement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Body mass index (BMI) between 25 and 45 kg/m2
* English speaking
* Have access to the Internet via a computer and smartphone compatible with Empower and Commercial Apps, and basic knowledge of how to use this technology.
* Agree to sharing of data entered in the Empower and Commercial Apps intervention systems.
* Agree to ShapeUp's privacy policy and user agreement.

Exclusion Criteria:

* Report health problems that make weight loss or unsupervised exercise unsafe or unreasonable
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Are currently pregnant or breastfeeding, or intend to become pregnant in the next 12 months
* Are planning to move outside of the greater Providence area within the next 12 months
* Report any cognitive or physical limitations that preclude use of a personal computer
* Have participated in a study conducted by the WCDRC in the past 2 years
* Have followed a commercial weight-loss program within the previous 6 months or who are currently following a commercial weight loss program
* Weight loss of ≥ 5% of initial body weight in the last 6 months
* History of clinically diagnosed eating disorder excluding Binge Eating Disorder.
* Previous surgical procedure for weight loss
* Currently taking weight loss medication\
* Treatment of cancer within the last 6 months
* Have any medical or psychological condition, or life situation, that would make participation in a weight loss program inadvisable in the opinion of the principal investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Body Weight (kg) | 6 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Resarch Center, Providence, Rhode Island, United States